CLINICAL TRIAL: NCT03165305
Title: The Role of Sustained Inflation on Short Term Respiratory Outcomes in Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Associate Professor, MD,PhD, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 123
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Distress Syndrome, Newborn; Transient Tachypnea of the Newborn; Respiratory Morbidity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Transient Tachypnea of the Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained Inflation Group (Experimental): Includes the infants who administered sustained inflation for 5 seconds with a pressure of 30cm H20 immediately after the delivery.
  Interventions: Other: Sustained Inflation
- No Intervention group (No Intervention): Includes routine neonatal care in the delivery room

INTERVENTIONS:
Other: Sustained Inflation — Administering a pressure of 30 cm H20 by a T-piece resuscitator for 5 seconds immediately after birth.
  Arms: Sustained Inflation Group

SUMMARY:
Sustained inflation (SI) has been reported to be effective for reducing the need for intubation and/or invasive ventilation in preterm infants. However, it has also an important role to support the initial breaths and liquid removal from the airways. Therefore, the investigators hypothesized that SI performed just after birth may help to facilitate the transitional period and decrease the incidence of early respiratory morbidities such as transient tachypnea in term infants.

ELIGIBILITY:
Inclusion Criteria:

* term newborns
* parental informed consent
* inborn infants

Exclusion Criteria:

* major congenital/chromosomal abnormalities
* lack of informed consent
* outborn infants
* Premature infants

Max Age: 2 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Morbidity | 2 hours
  RDS, TTN, requirement for supplemental oxygen, intubation or mechanical ventilation support

CONTACTS AND LOCATIONS:
Overall Officials: Merih Cetinkaya, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No